CLINICAL TRIAL: NCT04161482
Title: An Open Label Study to Evaluate the Impact of Duration of Subcutaneous Infusion of a Novel, pH Neutral Formulation of Furosemide (Furoscix®) on Safety and Local Skin Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Collaborators: Clinical Trial Data Services, Inc. (Unknown); CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: scP-01-007
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Healthy
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: The initial cohort (Cohort 1) will receive 80 mg (10 mL) with a bi-phasic delivery profile over 5 hours.
  Cohort 2a will evaluate a 2-hour infusion and Cohort 2b will be a bi-phasic delivery over 2 hours.
  Cohorts 3 and 4 will deliver the Furoscix over one hour and 30 minutes, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort One (Experimental): A bi-phasic delivery over 5 hours
  Interventions: Drug: Furosemide 80 mg (8 mg/mL)
- Cohort 2a (Experimental): Continuous infusion over 2 hours
  Interventions: Drug: Furosemide 80 mg (8 mg/mL)
- Cohort 2b (Experimental): Bi-phasic delivery over 2 hours
  Interventions: Drug: Furosemide 80 mg (8 mg/mL)
- Cohort 3 (Experimental): Continuous infusion over 1 hour.
  Interventions: Drug: Furosemide 80 mg (8 mg/mL)
- Cohort 4 (Experimental): Continuous infusion over 30 minutes.
  Interventions: Drug: Furosemide 80 mg (8 mg/mL)

INTERVENTIONS:
Drug: Furosemide 80 mg (8 mg/mL) — Furoscix will be administered as a subcutaneous infusion.

SUMMARY:
This is a Phase 1 study to evaluate the safety and tolerability of shortened subcutaneous infusions of Furoscix.

DETAILED DESCRIPTION:
Furoscix 80 mg will be administered as a subcutaneous infusion following a step-wise decrease in infusion times starting with a 5 hour infusion time. Subsequent cohorts will enroll following a safety assessment of the prior cohort. While maintaining the 80 mg dose, infusion time will ultimately be reduced to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion only if all of the following criteria are met:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Male and female Subjects 45-80 years of age.
3. Have the ability to understand the requirements of the study and is willing to comply with all study procedures.
4. In the opinion of the investigator, able to participate in the study.

Exclusion Criteria:

A Subject is not eligible for inclusion if any of the following criteria apply:

1. Receipt of loop diuretics (furosemide, bumetanide or torsemide) or thiazide diuretics (hydrochlorothiazide or metolazone) within 24 hours of study drug.
2. Receipt of potassium-sparing diuretics (spironolactone, amiloride) or oral calcium, potassium or magnesium supplements (including multi-vitamins) within 24 hours of study drug.
3. History of allergy to furosemide, sulfonamides or other loop diuretics.
4. Any skin conditions currently requiring medical therapy.
5. History of diabetes.
6. Presence or need for urinary catheterization, urinary tract abnormality or disorder interfering with urination.
7. Serum sodium <130 mEq/L at screening.
8. Serum potassium < 3.5 or > 5.5 mEq/L at screening.
9. Serum magnesium < 1.5 or > 2.5 mEq/L at screening.
10. Serum chloride < 96 or > 106 mEq/L at screening.
11. Serum calcium < 8.5 or > 10.5 mg/dL at screening.
12. Estimated Glomerular Filtration Rate (GFR) < 30 mL/min/1.73 m2 by simplified Modification of Diet in Renal Disease (sMDRD) equation at screening.
13. Systolic BP (SBP) < 90 mm Hg at screening or baseline.
14. Heart rate > 110 beats per minute (BPM) at screening or baseline.
15. History of tinnitus or hearing impairment, including deafness.
16. Temperature > 38°C (oral or equivalent) at screening or baseline.
17. Blood alcohol concentration > 2 mg/dL (0.02%) at screening or baseline.
18. Female Subject who is pregnant or lactating.
19. History of major abdominal surgery affecting the needle placement site.
20. History of benign prostatic hyperplasia (BPH), prostatitis or prostate cancer.
21. Urinary retention due to bladder emptying disorders and/or urethral narrowing.
22. History of liver disease, cirrhosis, or ascites.
23. Any local abdominal skin condition on the day of treatment i.e. sunburn, rash, eczema, etc.
24. Allergies and/or sensitivities to adhesive bandages or medical tape.
25. Any surgical or medical condition which in the opinion of the Investigator may interfere with participation in the study or which may affect the outcome of the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Infusion Site Pain (11 Point Pain Scale) | 8 hours
  Assessment of pain will be conducted upon placement of the subcutaneous (SC) needle, upon activation of SC infusion and periodically during the infusion and post-infusion completion for up to 8 hours after the start of the infusion using a standardized 11 point pain scale. Score will range from 0 to 10, where zero is equivalent to no pain and 10 is equivalent to the worst possible pain.

SECONDARY OUTCOMES:
Safety (Adverse Events) | Hours 1-8 and at the 24-48 hour follow up visit.
  Incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) will be assessed from the start of study drug administration through 24-48 hours after the start of the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Arora, MD, Principal Investigator — Aventiv Clinical Research
Locations (1):
- Aventiv Clinical Research, Columbus, Ohio, United States